CLINICAL TRIAL: NCT00327002
Title: A Mechanistic Study of the Effects of LY518674 on HDL C Metabolism
Brief Title: A Mechanistic Study of the Effects of LY518674 on High-Density Lipoprotein Cholesterol (HDL-C) Metabolism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 804137 PALMS; GCRC # 0995
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Metabolic Syndrome X
Keywords: Low HDL; Metabolic syndrome; low HDL Cholesterol in setting of metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — LY 518674

INTERVENTIONS:
Drug: LY518674

SUMMARY:
Agents that increase HDL-C via reverse cholesterol transport could provide a new therapeutic option for the prevention of atherosclerotic cardiovascular disease. The investigators propose to investigate the effects of LY518674 on components that may likely affect atherogenesis in patients with the metabolic syndrome including HDL-C metabolism and reverse cholesterol transport pathways, the inflammatory response, and oxidative stress in human subjects.

As an agonist of the nuclear peroxisome proliferator activated receptor (PPAR) alpha, LY518674 may affect the transcription of genes that encode various proteins involved in atherogenesis. This study will explore the consequences of altered transcription such as changes in messenger ribonucleic acid (mRNA) and protein levels as well as protein activity.

DETAILED DESCRIPTION:
Study Objectives

I. Primary Objective:

* To determine the effects of LY518674 on the Apo A-I production rate (calculated from the fractional synthetic rate and the fractional catabolic rate) in subjects with the metabolic syndrome and low HDL-C.

II. Secondary Objectives:

* To determine the effects of LY518674 on markers of reverse cholesterol transport by analyzing changes in serum cholesterol efflux capacity (an in vitro cell-based assay).
* To determine the effects of LY518674 on the activity of lecithin cholesterol acyltransferase (LCAT), cholesterol ester transfer protein (CETP), lipoprotein lipase, hepatic lipase, and endothelial lipase.
* To determine the effects of LY518674 on plasma lipids, lipid subfractions, free fatty acids, and the free fatty acid metabolite, beta-OH butyrate.
* To determine the effects of LY518674 on high-density lipoprotein (HDL), low-density lipoprotein (LDL) and very low-density lipoprotein (VLDL) particle size using nuclear magnetic resonance (NMR).
* To determine the effects of LY518674 on Apo A-II and Apo B-100 kinetics.
* To determine the effects of LY518674 on hsCRP.
* To determine the safety and tolerability of LY518674

Study Design:

Study H8D-MC-EMBG is a single site, randomized, placebo-controlled, double-blind, parallel study. A minimum of 40 subjects with low HDL cholesterol and metabolic syndrome will be randomized to receive double-blind administration of LY518674 100 mcg/day or placebo for 8 weeks. There is a safety visit every 2 weeks after treatment has been initiated, resulting in 7 visits over 10 weeks. There are 2 inpatient visits at zero and eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of > = 18 and < = 80.
2. HDL-C < 40 mg/dL in men; HDL-C < 50 mg/dL in women.
3. At least two of the following criteria ([a], [b], [c], or [d]) listed below:

   1. Abdominal obesity defined by waist circumference: non-Asian men > = 40 inches (102 cm) and non-Asian women > = 35 inches (88 cm); Asian men > = 35 inches (88 cm) and Asian women > = 31 inches (79 cm),
   2. Blood pressure > = 130 systolic, or > = 85 diastolic mm Hg (on average of 3 measurements) in untreated patients OR if patient is taking > = 1 approved anti-hypertensive agent,
   3. Fasting glucose > = 100 mg/dL and < 126 mg/dL,
   4. Fasting triglycerides > 150 mg/dL and < 600 mg/dL.
4. Have given signed informed consent to participate in the study.
5. Women of child-bearing potential, that is, women not surgically sterilized and between menarche and 1 year post menopause, must test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control (for example, use of oral contraceptives or Norplant®; a reliable barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices]; partner with vasectomy; or abstinence) during the study and for one month following the last dose of study drug.
6. Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

Potential study subjects may not be entered into the study if any of the following apply:

1. Lipid-altering medications that meet any of the following criteria prior to the screening visit, are planned or are likely to be required during the course of the study:

   1. Subjects who have not been on a stable dose of statin therapy within 4 weeks.
   2. Subjects who have received fish oil dietary supplements > 2 g/d within 4 weeks.
   3. Use of more than 250 mg per day of niacin within 6 weeks; fibrates within 12 weeks; or thiazolidinediones (TZDs) within 12 weeks.
   4. Orlistat and bile acid sequestrants are not permitted within 4 weeks.
   5. Ezetimibe is not permitted within 4 weeks.
   6. Postmenopausal women who have not been on a stable selective estrogen receptor modulator (SERM) dose within 4 weeks.
2. Investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
3. Lilly employees.
4. Within 30 days of the initial dose of study drug, have received treatment with a drug that has not received regulatory approval for any indication.
5. Have previously completed or withdrawn from this study or any other study investigating LY518674.
6. Patients with diabetes or receiving PPARs consisting of gamma, alpha, delta agonists or gamma, alpha, delta antagonists, or partial agonists alone and in any combination.
7. Uncontrolled hypertension defined as systolic blood pressure > 180 mm Hg, diastolic blood pressure > 100 mm Hg.
8. Have a serum creatinine > = 2 mg/dL, or nephrotic syndrome, end stage renal disease and use renal replacement therapy such as hemodialysis or peritoneal dialysis.
9. Liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP] or total bilirubin) > 1.5 x the upper limit of normal (ULN).
10. Have hemoglobin < 10.5 gm/dL in women and < 11.5 gm/dL in men.
11. Have or have had any clinical manifestations of coronary heart disease (CHD) such as unstable angina, acute coronary syndrome, a myocardial infarction (MI), a coronary revascularization procedure including stent placement, or any other condition for which statin therapy is recommended for secondary prevention of cardiovascular disease as seen in type 1 and 2 diabetes mellitus or genetic forms of hypercholesterolemia (for example, familial hypercholesterolemia).
12. History of congestive heart failure (CHF).
13. History of a non-skin malignancy within the previous 5 years.
14. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition.
15. Surgery in the last 30 days, or have planned or are likely to require major surgery during the course of the study.
16. Subject-reported history of human immunodeficiency virus infection.
17. Have chronic alcohol or drug abuse.
18. Subjects who have an average weekly alcohol intake that exceeds 14 units per week (1 unit = 12 oz of beer; 5 oz of wine; 1.0 oz of distilled spirits).
19. Have any other medical condition, laboratory abnormality, or circumstance prior to randomization, which, in the opinion of the investigator, could affect subject safety, preclude evaluation of response, or prohibit the ability to comply with study procedures or completion of the study.
20. Known allergies to LY518674 or related compounds.
21. Known allergies to deuterated leucine or related compounds.
22. Have a history of hypersensitivity or intolerance to drug preparations containing PPAR alpha agonists such as clofibrate (example: Atromid-S®), fenofibrate (examples: Tricor® or Lofibra®), or gemfibrozil (example: Lopid®).
23. An abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risk of participating in the study, such as a corrected QT interval > 450 msec for men and > 470 msec for women.
24. Have or have had a history of a chronic muscular or neuromuscular disease including a history of prior rhabdomyolysis or drug-induced myopathy (for example, statin or fibric acid), or an unexplained elevation in creatine kinase (CK) > = 3 x ULN.
25. Cardiac troponin I level at or above the lower limit of detection at entry, with the lower limit of detection being defined by the performing reference laboratory.
26. Have a history of symptomatic postural hypotension or postural dizziness.
27. Are currently using, have used within 2 months prior to screening visit, plan to use or are likely to require during the course of the study drugs, herbal preparations, or foods that may inhibit or induce cytochrome P450 3A.
28. Have thyroid-stimulating hormone (TSH) levels outside normal reference range for the central laboratory. Subjects who are clinically euthyroid and on stable thyroid replacement therapy for 2 months prior to screening and who are anticipated to remain on this dose throughout the trial period are acceptable exceptions to this criterion.
29. Currently adhering to, have used within 2 months prior to screening, or have plans to adopt diets with aggressive carbohydrate restrictions for weight loss, such as but not limited to Atkins or South Beach diets.
30. Currently use, have used within 2 months prior to screening, or plan to use during the trial period dietary supplements or over the counter formulations intended for weight loss.
31. Have active hepatobiliary disease, serologic evidence of past or active hepatitis B or C, OR past or active gallbladder disease.
32. Use any immunosuppressive therapy within 2 months prior to screening or are likely to require immunosuppressive therapy during the course of the study.
33. Subjects requiring hormone therapy using glucocorticoids within 2 to 3 months prior to study entry (topical preparations, nasal and intra-articular administration, as well as physiologic replacement for Addison's disease or hypopituitarism are permitted).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rader, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- John Millar, Philadelphia, Pennsylvania, United States